CLINICAL TRIAL: NCT01979380
Title: A Randomized, Double-blind, Placebo-controlled, Ascending Single Oral Dose, Phase I Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetics of KD101 in Healthy Male Subjects
Brief Title: Phase I Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetics of KD101 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kwang Dong Pharmaceutical co., ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: KD101-101
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Drug Toxicity
Keywords: KD101; Anti-obesity Agents
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KD101 (Experimental)
  Interventions: Drug: KD101
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: KD101 — 200mg (1casule), 600mg (3 capsule), 1000mg (5 capsule), 1400mg (7 capsule) PO, once in the morning
  Other Names: KD101 soft capsule 200mg
  Arms: KD101
Drug: placebo — PO, once in the morning
  Other Names: KD101 placebo
  Arms: placebo

SUMMARY:
To Evaluate the safety and tolerability after KD101 single oral dosing in healthy male subjects

To Evaluate the pharmacokinetic property after KD101 single oral dosing in healthy male subjects

To Evaluate the effect of food on bioavailability after KD101 single oral dosing in healthy male subjects

DETAILED DESCRIPTION:
This clinical trial is a dose block-randomized, double-blinded, placebo controlled, single ascending dose, food interaction study. AEs, PE, Vital signs, ECGs and clinical lab tests will be assessed to evaluate the safety and tolerability, and blood and urine will be collected to evaluate the pharmacokinetic parameters.

This single ascending dose, food interaction study will be conducted with the KD101 dose of 200, 600, 1000 and 1400 mg. After evaluating the safety and pharmacokinetic parameters in the single dose KD101 group of 200mg, next higher dose of KD101 will be administered and evaluated and food interaction will be evaluated in the KD101 group of 600mg.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who listened the properties of this clinical trial and signed IRB approved-ICF by voluntary consent
* Male adults aged 20 to 55 years at screening
* Healthy volunteer whose BMI ≥ 18
* Subjects who are adequate to this trial by physical examination, lab examination, diagnosis from physician

Exclusion Criteria:

* Subjects who had clinically significant disease history (liver,kidney,nervous,pulmonary,endocrinal,urinary,cardiovascular,musculoskeletal,mental system,blood,tumor) or diagnosed within 1 month from screening
* Subjects who had gastrointestinal disease(Crohn's disease, ulcer, acute/chronic pancreatitis) that affect the absorption of test drug or gastrointestinal operation (However, appendectomy, herniotomy induced by acute appendicitis are excluded)
* Subjects who had / or were suspected to had following history. [myocardial infarction (diagnosed by cardiac enzyme and/or diagnostic ECG), cerebral infarction/stroke , arrhythmia needed to medical treatment, unstable angina, pulmonary hypertension]
* Subjects who had positive result to Human Immunodeficiency Virus, Hepatitis B virus, Hepatitis C virus during screening
* Subjects who had allergy history (ex. allergy for aspirin, antibiotics, etc) or had clinically-significant allergy
* Subjects whose systolic BP was <85mmHg or >145mmHg, or diastolic BP was <50mmHg or >95mmHg, or pulse was >100/min after 3 minute-seating position. (BP can be re-measured twice at leat 5 minute-interval)
* Subjects who would take prescribed/oriental drug(within 2 weeks from the first dosing day) or OTC drug or vitamines (within 1 weeks from the first dosing day)
* Subjects who drink over than 21 unit (1 unit = 10g of pure alcohol) or cannot quit drinking alcohol during clinical trial period
* Subjects who ate following food within 2 days from the first dosing day or cannot quit following food [grapefruit-contain food, caffein-contain food(coffee, green tea, black tea, soft drink, coffee milk, energy drink)]
* Subjects who didn't agree contraception
* Subjects who didn't agree to quit smoke
* Subjects who donated his/her blood within 2 months (whole blood) / 1 month (apheresis) or who took transfusion within 1 month
* Subjects who participated another clinical trials within 3 months from first dosing day. (The clinical trial completion day is defined as the last dosing day of past clinical trial)
* Subjects who are not adequate to this trial by lab examination and another reason

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Cmax, AUClast, AUCinf, Tmax, t1/2, fe, CL/F, Vd/F, % AUCextra, CLR | single dose

CONTACTS AND LOCATIONS:
Overall Officials: Howard Lee, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea